CLINICAL TRIAL: NCT00464698
Title: Duloxetine for the Treatment of Obsessive Compulsive Disorder
Brief Title: Duloxetine for the Treatment of Obsessive Compulsive Disorder (OCD)
Acronym: FIJ-MC-1003
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Darin Dougherty, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-002159; FIJ-MC-1003
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; Obsessive Compulsive Disorder; Obsessions; Compulsions; Duloxetine; Cymbalta
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Obsessive Behavior; Compulsive Behavior | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Study Participants (Experimental): Duloxetine 30mg: Dose level 1 (Week 1) Duloxetine 60mg: Dose level 2 (Wks 2-4) Duloxetine 120mg: Dose level 3 (Wks 3-7)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Participants received increasing amounts of Duloxetine for 7 weeks.
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to assess the efficacy of Duloxetine in the treatment of obsessive compulsive disorder.

DETAILED DESCRIPTION:
Obsessive compulsive disorder affects approximately 3% of the population. Treatment options include the selective serotonin reuptake inhibitors (SSRIs), dual serotonin and norepinephrine reuptake inhibitors (SNRIs), and behavioral therapy. Duloxetine is a new SNRI. This study aims to assess the efficacy of duloxetine for the treatment of OCD.

Before subjects give written informed consent, they are made aware of alternatives to participation in this study, which can include independently seeking pharmacotherapy or cognitive behavioral treatment for OCD. Patients will then begin open-label treatment with duloxetine at 30 mg/day and will be seen again in one week (Visit 2). At Visit 2, patients will be assessed and, if they are not experiencing any significant side effects, the dose will be increased to 60 mg/day. Patients who are experiencing significant side effects at 30 mg/day will be discontinued from the study and offered standard treatment in our clinic. Patients taking 60 mg/day will then return for assessment in four weeks (Visit 3). At this time, if they are not experiencing any significant side effects, the dose will then be increased to 120 mg/day. Patients who are unable to tolerate 120 mg/day will have their dose decreased back down to 60 mg/day and will continue the trial. End of study final statistical analyses will be conducted both including and excluding these patients. Remaining assessments will be every 4 weeks (Visits 4, 5, 6). Thus, in total this is a 17-week study with 12 weeks at the high dose believed to be necessary for response.

At each visit following the initial visit, patients will be assessed using the Y-BOCS, BDI, BAI, and CGI. The Q-LES-Q will only be administered at the initial and last visit.

The study procedure is similar to standard medical treatment for OCD at MGH. Like standard care, participants start on the lowest dose of the medication and then increase that dose to the maximally tolerated level. Barring any significant side effects, the patient remains on that dose for 4-8 weeks to provide the medication with an adequate trial period. At the end of that period, efficacy would be assessed and other alternatives would be discussed.

One difference between the study and standard care is that the study will provide more assessment through verbal and written scales. This additional assessment could greatly benefit the patient as they decide between other treatment options. Another difference is that participants cannot be involved in current behavior therapy throughout the study. Many patients choose to pursue medical treatment without behavior therapy in standard care; however, in standard care, they have the option of pursuing both concurrently or pursuing just behavior therapy. If a patient wishes to pursue just behavior therapy or receive medication and therapy concurrently, then other forms of treatment at MGH might be more appropriate. If they only want medical treatment, the study is similar to standard care at a lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD by DSM-IV
* Age 18-65
* Y-BOCS greater than 20
* Written informed consent
* Females of childbearing potential must have a negative serum or urinary beta-HCG test.

Exclusion Criteria:

* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception.
* Patients who, in the investigator's judgment, pose a serious suicidal or homicidal risk.
* Serious or unstable medical illness including cardiovascular (including hypertension), hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease. Patients on anticoagulant therapy.
* History of seizure disorder
* Comorbid bipolar disorder, psychosis, organic mental disorder, or developmental disorder
* If there is a history of substance abuse, patients in remission at least 6 months.
* Currently being treated with behavioral therapy, specifically exposure and response prevention, for OCD.
* Other medications for medical disorders that may interfere with duloxetine
* Current major depression or prescribed an antidepressant for major depression within the past 12 months. We will assess depressive symptoms with the BDI throughout the course of the study in order to assess subsyndromal depressive symptoms and to assess for the emergence of depressive symptoms.
* Taken other psychotropic medication within 2 weeks of beginning the study (4 weeks for fluoxetine).
* More than 1 adequate trial (at least 10 weeks at maximally tolerated dose) with another SSRI in the past.
* Known hypersensitivity to duloxetine or any of the inactive ingredients.
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or potential need to use an MAOI drug during the study or within 5 days of discontinuation of study drug.
* Patients with uncontrolled narrow-angle glaucoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darin D Dougherty, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dougherty DD, Corse AK, Chou T, Duffy A, Arulpragasam AR, Deckersbach T, Jenike MA, Keuthen NJ. Open-label study of duloxetine for the treatment of obsessive-compulsive disorder. Int J Neuropsychopharmacol. 2015 Jan 30;18(2):pyu062. doi: 10.1093/ijnp/pyu062. Print 2015. PMID 25637377
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pubmed/25637377

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Duloxetine Week 1 dose: 30mg Duloxetine Weeks 2-4 dose: 60mg Duloxetine Weeks 5-17 dose: 120mg
Period: Period 1: 30 mg
Arm/Group | All Study Participants
Started | 20
Completed | 17
Not Completed | 3
Period: Period 2: 60 mg
Arm/Group | All Study Participants
Started | 17
Completed | 17
Not Completed | 0
Period: Period 3: 120mg
Arm/Group | All Study Participants
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine: Duloxetine: Week 1 dose: 30mg, Weeks 2-4 dose: 60mg, Weeks 5-17 dose: 120mg
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.90 (10.66)
Age, Customized [Mean (Standard Deviation); unit: years] — Age of OCD onset
  years
    Age of OCD onset | 15.35 (10.479)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
Yale-Brown Obsessive Compulsive Scale (YBOCS) [Mean (Standard Deviation); unit: units on a scale] — Minimum score possible: 0 Maximum score possible: 40
  Greater scores indicate higher symptom severity
  units on a scale | 27.45 (4.08)
Duration of illness [Mean (Standard Deviation); unit: years] — Mean duration of OCD
  years | 14.80 (12.88)

OUTCOME MEASURES:

1. Primary Outcome: Y-BOCS Scores at 1st and Last Visit
Description: OCD symptom change. This is the intention-to-treat analyses (with all 20 subjects included) rather than just the subjects who completed the treatment.
Time Frame: Week 0 to 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
units on a scale
  Baseline YBOCS score | 27.45 (4.08)
  Final YBOCS score | 20.45 (7.57)

2. Secondary Outcome: BDI (Beck Depression Inventory) - First and Last Visit (Week 0 and Week 17).
Description: Depression severity, such that higher scores on the BDI are reflective of more severe depression.
  BDI minimum score: 0 MDI maximum score: 63
Time Frame: Week 0 to 17
Population: 20 participants with OCD were enrolled in a 17-week, open label treatment trial with duloxetine.
Measure: Mean (Standard Deviation); unit: units on a self-report questionnaire
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
units on a self-report questionnaire
  Baseline BDI (Week 0) | 10.30 (6.98)
  Final Visit BDI (Week 17) | 6.95 (6.10)

3. Secondary Outcome: BAI (Beck Anxiety Inventory) - First and Last Visit (Week 0 and Week 17)
Description: Anxiety severity, such that a higher score on the BAI reflects more severe anxiety.
  Minimum value: 0 Maximum value: 63
Time Frame: Week 0 to 17
Population: 20 participants with OCD were enrolled in a 17-week, open label treatment trial with duloxetine.
Measure: Mean (Standard Deviation); unit: units on a self-report questionnaire
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
units on a self-report questionnaire
  Baseline BAI (Week 0) | 10.70 (11.54)
  Final Visit BAI (Week 17) | 6.75 (7.05)

4. Secondary Outcome: QLESQ (Quality of Life, Enjoyment, and Satisfaction Questionnaire) - First and Last Visit (Week 0 and Week 17)
Description: Quality of life, such that lower score reflects poorer quality of life
  Minimum score: 16 Maximum score: 80
Time Frame: Week 0 to 17
Population: 20 participants with OCD were enrolled in a 17-week, open label treatment trial with duloxetine.
Measure: Mean (Standard Deviation); unit: units on a self-report questionnaire
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
units on a self-report questionnaire
  Baseline Q-LES-Q (Week 0) | 70.14 (14.03)
  Final Visit Q-LES-Q (Week 17) | 74.55 (12.03)

5. Secondary Outcome: Clinical Global Impressions Scale at Week 3 and Week 17
Description: Global severity of illness, such that a higher score reflects worse global severity
  Minimum score: 2 Maximum score: 14
Time Frame: Week 3 to 17
Population: 20 participants with OCD were enrolled in a 17-week, open label treatment trial with duloxetine.
Measure: Mean (Standard Deviation); unit: units on a self-report questionnaire
Arm/Group | Duloxetine
Number analyzed (Participants) | 20
units on a self-report questionnaire
  Baseline CGI (Week 3) | 4.0 (0)
  Final Visit CGI (Week 17) | 2.70 (.923)

ADVERSE EVENTS:
Arm/Group | Duloxetine: Week 1 Dose: 30mg | Duloxetine Weeks 2-4 Dose: 60mg | Duloxetine Weeks 5-17 Dose: 120mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 10/20 | 7/17 | 7/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine: Week 1 Dose: 30mg (N=20) | Duloxetine Weeks 2-4 Dose: 60mg (N=17) | Duloxetine Weeks 5-17 Dose: 120mg (N=14)
nausea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 4 (4)
fatigue (General disorders) | 5 (5) | 5 (5) | 6 (6)
sexual dysfunction (Reproductive system and breast disorders) | 2 (2) | 4 (4) | 3 (3)
headache (General disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No